CLINICAL TRIAL: NCT00051454
Title: A Randomised, Placebo-Controlled, Double-Blind, Phase I/IIa Clinical Trial to Evaluate the Safety and Immunogenicity of a Candidate Prophylactic DNA Prime-rFPV Boost HIV Vaccination Strategy
Brief Title: Evaluation of the Safety of and Immune Response to an HIV Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N01-AI05395
Record Dates: First submitted 2003-01-10; First posted 2003-01-13 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: HIV DNA plasmid vaccine plus recombinant fowlpox vector

SUMMARY:
This study will examine the safety and immune response to a two-part HIV vaccine. Healthy volunteers who are at low risk of HIV infection will receive either active vaccine or a placebo.

DETAILED DESCRIPTION:
The purpose of this study is to examine the safety and immunogenicity of a candidate vaccine strategy for HIV prophylaxis using a DNA-prime plus recombinant fowlpox boost. The DNA plasmid and fowlpox vector contain HIV genes. However, these vaccines contain only some HIV genes and cannot themselves cause HIV or AIDS.

Eligible volunteers at low risk of HIV infection will be randomized to receive either active vaccine or placebo injections at Day 0, Week 4, and Week 8. Intensive immunologic and safety monitoring will be done during the first 16 weeks of the study. Follow-up will continue to Week 52.

ELIGIBILITY:
Inclusion Criteria

* HIV negative.
* Acceptable methods of contraception.

Exclusion Criteria

* Identifiable risk behavior for HIV infection, including: sexual partners of HIV positive people, sexual intercourse with a partner of unknown HIV status if that partner is reported to be at higher risk for HIV infection, gay men reporting any unprotected anal intercourse with partners of unknown status in the 12 months preceding study entry, individuals diagnosed with a sexually transmissible infection (STI) in the 12 months preceding entry that may have been acquired through anal or vaginal intercourse, individuals reporting sharing of injecting equipment in the last 12 months.
* HIV candidate vaccines in a previous HIV vaccine trial.
* Live attenuated vaccines within 60 days prior to entering the study. Whole killed, toxoid, or sub-unit vaccines (e.g., influenza, pneumococcal, tetanus, and hepatitis B) are not exclusionary within 4 weeks prior to the scheduled experimental HIV vaccines.
* Hypersensitivity to egg products or a known history of anaphylaxis or any other serious adverse reactions to vaccination.
* History of serious allergic reaction requiring hospitalization or emergency medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension) to any substance.
* Significant illness requiring immunomodulatory or cytotoxic therapy.
* History of cancer unless there is evidence of surgical excision followed by a sufficient observation period to give a reasonable assurance of cure.
* Blood products or immunoglobulins within 6 months prior to entering the study.
* Experimental or investigational agents within 30 days prior to entering the study.
* Recreational and/or therapeutic drug use that might compromise the study participant's safety.
* Medical or psychiatric condition or occupational responsibilities that preclude compliance with the protocol.
* Pregnant or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2003-03; Study Completion 2005-02

PRIMARY OUTCOMES:
Safety and adverse events among the two vaccination groups
lymphoproliferative (LP) responses to HIV antigens, as assessed by LP assays at Week 9
CD8+ T cell responses to HIV antigens, as assessed by ELIspot assay of interferon gamma (IFN-g) secreting cells at Week 9

SECONDARY OUTCOMES:
Proportion of patients with positive LP assay and ELISPOT assay responses
intracellular cytokine staining (ICS) of IFN-g/CD69 and flow cytometry
51-Cr release cytotoxic T cell lymphocyte assay
HLA class I tetramer analyses
anti-HIV gag, pol and env antibodies, as assessed by ELISA and Western blot
behavioral changes in study participants

CONTACTS AND LOCATIONS:
Overall Officials: David A Cooper, MD, DSc, Study Director — National Centre in HIV Epidemiology and Clinical Research, University of New South Wales
Locations (1):
- National Centre in HIV Epidemiology and Clinical Research, Sydney, New South Wales, Australia

REFERENCES:
- [Result] Kelleher AD, Puls RL, Bebbington M, Boyle D, Ffrench R, Kent SJ, Kippax S, Purcell DF, Thomson S, Wand H, Cooper DA, Emery S. A randomized, placebo-controlled phase I trial of DNA prime, recombinant fowlpox virus boost prophylactic vaccine for HIV-1. AIDS. 2006 Jan 9;20(2):294-7. doi: 10.1097/01.aids.0000199819.40079.e9. PMID 16511428
- See also: Related Info — http://www.med.unsw.edu.au/nchecr